CLINICAL TRIAL: NCT04446377
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Study of LAM-002A for the Prevention of Progression of COVID-19
Brief Title: A Study of LAM-002A for the Prevention of Progression of COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OrphAI Therapeutics (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAM-002A-CVD-CLN01
Record Dates: First submitted 2020-06-23; First posted 2020-06-24 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: COVID-19 Disease
Keywords: COVID-19; SARS-CoV-2; Apilimod Dimesylate; LAM-002A; Coronavirus; AI Therapeutics
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — apilimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LAM-002A (Experimental): LAM-002A (Apilimod Dimesylate) 125mg in five 25-mg capsules BID for 10 days
  Interventions: Drug: Apilimod Dimesylate Capsule
- Placebo (Placebo Comparator): (microcrystalline cellulose) in 5 capsules BID for 10 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Apilimod Dimesylate Capsule — LAM-002A is formulated in capsules containing 25 mg of apilimod dimesylate. The capsule is Swedish orange, Size 0.
  Arms: LAM-002A
Other: Placebo — Microcrystalline cellulose in Swedish orange, Size 0 capsules
  Arms: Placebo

SUMMARY:
This is a clinical trial to evaluate the efficacy of LAM-002A compared to placebo treatment in adults with a confirmed SARS-CoV-2 infection who are receiving standards supportive care in an outpatient setting.

DETAILED DESCRIPTION:
This is a Phase II randomized, double-blind, placebo-controlled, clinical study to evaluate the efficacy of LAM-002A compared to placebo treatment in adults with a confirmed SARS-CoV-2 infection who are receiving standard supportive care in an outpatient setting.

Study eligibility will be assessed during screening. All study participants must sign a written informed consent and satisfy the inclusion and exclusion criteria for the study. Confirmation of SARS-CoV-2 infection, medical history, and current medication will be assessed for each consenting participant at screening.

Study participants will be randomized in a 1:1 ratio, to receive study therapy (either LAM-002A, 125 mg [5 capsules/dose]) PO BID or placebo [5 capsules/dose] PO BID) for 10 days. Participants who experience an adverse event (AE) considered to be related to study therapy may have a decrease in study dose of LAM-002A to 100 mg [4 capsules/dose]) PO BID or placebo [4 capsules/dose] PO BID). After the start of treatment on Day 1, participants will be followed at Days 4,6,8,11,22, and 28. Days 6,8, and 22 will be phone visits. Participants can withdraw from the study therapy or study participation at any time.

The study will incorporate an interim safety analysis after the first 30 participants (15 on LAM-002A and 15 on placebo) have completed treatment and have been followed up for 11 days post-first dose. Recruitment and randomization will continue while this analysis is conducted. Recommendations from an independent Data Safety Monitoring Board (DSMB) will be used for decisions of early termination or study design adaptations.

Non-parametric and parametric statistical analysis will be conducted, as appropriate. For the comparison of the LAM-002A active arm and the control arm for the primary endpoint and secondary endpoints of drug effect, appropriate methods will be employed. Baseline subject characteristics, study therapy administration/compliance, safety, supportive care administration, and pharmacokinetics will be analyzed descriptively.

ELIGIBILITY:
Inclusion Criteria:

1. Written documentation of SARS-CoV-2 infection confirmed by a validated test.
2. Presence of greater than or equal to ≥1 of the following COVID-19-related symptoms indicating mild disease: fever (temperature ≥100.4), anosmia (loss of taste or smell), cough, sore throat, gastrointestinal complaints (e.g. nausea, vomiting, or diarrhea), chills, congestion, or runny nose, headaches, muscle or body aches, fatigue, or asymptomatic patients who have tested positive for COVID-19 via a validated test within the past 4 days.
3. If symptomatic, symptom onset less than or equal to ≤ 8 days.
4. For female participants of childbearing potential, a negative urine (or serum) pregnancy test.
5. For female participants of childbearing potential, willingness to use a protocol-recommended method of contraception from the start of the screening period until greater than or equal to ≥30 days after the final dose of study therapy. Note: A female subject is considered to be of childbearing potential unless she has had a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy; has medically documented ovarian failure (with serum estradiol and follicle-stimulating hormone [FSH] levels within the institutional laboratory postmenopausal range and a negative serum or urine beta human chorionic gonadotropin [βHCG]); or is menopausal (age ≥50 years with amenorrhea for ≥6 months).
6. For male participants who can father a child and are having intercourse with females of childbearing potential who are not using adequate contraception, willingness to use a protocol-recommended method of contraception from the start of study therapy until ≥30 days after the final dose of study therapy and to refrain from sperm donation from the start of study therapy until ≥90 days after administration of the final dose of study therapy. Note: A male subject is considered able to father a child unless he has had a bilateral vasectomy with documented aspermia or a bilateral orchiectomy.
7. Willingness and ability of the participant to ingest study drug capsules.
8. Willingness of the participant to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, study procedures, and study restrictions.
9. Evidence of a personally signed informed consent indicating that the participant is aware of the nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.

Exclusion Criteria:

1. Respiratory rate greater than or equal to ≥20 breaths per minute.
2. Oxygen saturation by pulse oximetry less than or equal to ≤93 percent % on room air or requirement for supplemental oxygen to maintain oxygen saturation greater than >93 percent %.
3. Total NEWS score greater than or equal to ≥6 or presence of a score of 3 on any of the individual NEWS parameters.
4. Radiographic evidence of pulmonary infiltrates (clinical X-ray within 2 days of referral)
5. Hepatic profile showing any of the following:

   * Serum alanine aminotransferase (ALT) greater than >5 × upper limit of normal (ULN) (CTCAE Grade greater than or equal to ≥3).
   * Serum aspartate aminotransferase (AST) greater than >5 × ULN (CTCAE Grade greater than or equal to ≥3).
   * Serum bilirubin greater than >1.5 × ULN (CTCAE Grade greater than or equal to ≥2).
6. Renal profile showing an estimated creatinine clearance (eClCR) less than <30 mL/minute (with eClCR to be calculated by the method at the laboratory performing the serum creatinine test).
7. Presence of a cancer with disease manifestations or therapy that could adversely affect subject safety or longevity, create the potential for drug-drug interactions, or compromise the interpretation of study results.
8. Significant cardiovascular disease (e.g. myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 1 month prior to start of study therapy; unstable angina; symptomatic peripheral vascular disease; CTCAE Grade greater than or equal to ≥2 congestive heart failure; or uncontrolled CTCAE Grade greater than or equal to ≥3 hypertension (diastolic blood pressure greater than or equal to ≥100 mmHg or systolic blood pressure greater than or equal to ≥160 mmHg) despite antihypertensive therapy.
9. Significant screening ECG abnormalities, including atrial fibrillation/flutter, 2nd degree atrioventricular (AV) block type II, 3rd-degree AV block, Grade greater than or equal to ≥2 bradycardia, or corrected QT (QTc by Fridericia [QTcF]) greater than >480 msec (Grade greater than >1).
10. Gastrointestinal disease (e.g. gastric or intestinal bypass surgery, pancreatic enzyme insufficiency, malabsorption syndrome, symptomatic inflammatory bowel disease, chronic diarrheal illness, bowel obstruction) that might interfere with drug absorption or with interpretation of gastrointestinal AEs.
11. Pregnancy or breastfeeding.
12. Prior solid organ transplantation.
13. Use within 5 days prior to randomization of an approved or investigational therapy intended to treat COVID-19 (e.g. remdesivir, , anti-interleukin [IL]-6 antibodies, therapeutic anti-SARS CoV-2 antibodies or post-convalescent plasma, anti- SARS CoV-2 vaccine, Bruton tyrosine kinase [BTK] inhibitor), use within 3 months of chloroquine or hydroxychloroquine. Note: participants are not precluded from undergoing evaluations involving observation, noninvasive diagnostic procedures or sampling, or questionnaires as follow-up to a prior study or as components of a concurrent noninterventional study.
14. Use within 5 days prior to randomization of a strong inhibitor or inducer of cytochrome P450 (CYP) 3A4 or expected requirement for chronic use of a strong inhibitor or inducer of CYP3A4 during study therapy.
15. Use within 5 days prior to randomization of drug that is a moderate-to-strong substrate of CYP2C9 (including warfarin, tolbutamide, phenytoin, glimepiride) or expected requirement for chronic use of such drugs during study therapy.
16. Use within 5 days prior to randomization of a drug known to prolong the QT interval
17. Ongoing immunosuppressive therapy including systemic or enteric corticosteroids. (Note: At study entry, participants may be using intraarticular, inhaled, or topical corticosteroids. During study therapy, participants may use systemic, enteric, intraarticular, inhaled, or topical corticosteroids as required for intercurrent conditions.)
18. Any illness, medical condition, organ system dysfunction, or social situation, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a participant's ability to provide informed consent, adversely affect the participant's ability to cooperate and participate in the study, or compromise the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar P, Mathayan M, Smieszek SP, Przychodzen BP, Koprivica V, Birznieks G, Polymeropoulos MH, Prabhakar BS. Identification of potential COVID-19 treatment compounds which inhibit SARS Cov2 prototypic, Delta and Omicron variant infection. Virology. 2022 Jul;572:64-71. doi: 10.1016/j.virol.2022.05.004. Epub 2022 May 16. PMID 35598394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by 8 investigators located at medical centers throughout the United States
Pre-assignment Details: The screening and baseline visits could occur on the same day. Day 1 of the study was the day the participant took the first dose of study drug after randomization.
Groups:
- LAM-002A: 71 participants were allocated to receive LAM-002A (Apilimod Dimesylate) 125 mg in five 25-mg capsules twice a day (BID) for 10 days.
  Participants were to be followed for 28 days from the start of LAM-002A treatment.
- Placebo: 71 participants were allocated to receive Placebo (microcrystalline cellulose) in 5 capsules BID for 10 days.
  Participants were to be followed for 28 days from the start of Placebo treatment.
Period: Overall Study
Arm/Group | LAM-002A | Placebo
Started | 71 | 71
Completed | 64 | 66
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Not eligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population included all participants randomized according to their initial randomized assignment regardless of the treatment actually received.
Groups:
- LAM-002A: 71 subjects were allocated to receive LAM-002A (Apilimod Dimesylate) 125 mg in five 25-mg capsules BID for 10 days.
- Placebo: 71 subjects were allocated to receive Placebo (microcrystalline cellulose) in 5 capsules BID for 10 days.
- Total: Total of all reporting groups
Arm/Group | LAM-002A | Placebo | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Continuous [Median (Full Range); unit: years] | 42.8 [18.7 to 70.4] | 43.3 [18.5 to 65.7] | 43.1 [18.5 to 70.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 34 | 34 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 27 | 52
  Not Hispanic or Latino | 45 | 44 | 89
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Patient Race: White | 64 | 61 | 125
  Patient Race: Black or African American | 2 | 7 | 9
  Patient Race: Asian | 3 | 0 | 3
  Patient Race: Other | 0 | 1 | 1
  Patient Race: Unknown | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 71 | 71 | 142
ECOG Performance Status [Count of Participants; unit: Participants]
  0: Fully active | 55 | 59 | 114
  1: Restricted | 16 | 11 | 27
  2: Ambulatory | 0 | 1 | 1
Oxygen Saturation [Median (Full Range); unit: percent] | 98.0 [95.0 to 100.0] | 98.0 [95.0 to 100.0] | 98.0 [95.0 to 100.0]
Temperature [Median (Full Range); unit: degrees Celsius] | 36.8 [35.7 to 38.6] | 36.8 [35.6 to 38.0] | 36.8 [35.6 to 38.6]

OUTCOME MEASURES:

1. Primary Outcome: Viral Load Change
Description: The primary efficacy outcome measure evaluated change in SARS-CoV-2 viral load at Day 4 from Day 1, of LAM-002A or placebo-treated participants. SARS-CoV-2 viral load was measured by a real-time quantitative reverse transcription polymerase chain reaction (qRT-PCR) test of nasopharyngeal samples. Analysis focused on log10 viral load on Day 4 compared to baseline viral load at Day 1 in participants with baseline viral load >100,000 copies/mL
Time Frame: 4 Days
Population: Antiviral efficacy population comprising of participants with baseline viral load >100,000 copies/mL = log10 viral load >5)
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- LAM-002A: 71 participants were allocated to receive LAM-002A (Apilimod Dimesylate) 125 mg in five 25-mg capsules BID for 10 days.
- Placebo: 71 participants were allocated to receive Placebo (microcrystalline cellulose) in 5 capsules BID for 10 days.
Arm/Group | LAM-002A | Placebo
Number analyzed (Participants) | 43 | 35
log10 copies/mL | -2.50 (2.35) | -1.99 (1.71)
Statistical Analysis 1: Comparison: LAM-002A vs Placebo; The analysis tested whether the viral load in nasopharyngeal samples was lower at Day 4 in those receiving LAM-002A compared to Placebo; Test type: Superiority — The alternative hypothesis for the statistical testing was that LAM-002A would induce greater changes in viral load from Day 1 to Day 4 than would Placebo; p = 0.35, Mixed Models Analysis — Pre-specified 2-sided significance level of 0.20; ANCOVA linear mixed model to evaluate the relative differences between the LAM-002A and Placebo groups in the log10 viral load from Day 1 to Day 4; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.47 to 0.53], Standard Error of Mean 0.51 — The difference between the groups (LAM-002A vs Placebo)

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: The number and percentage of LAM 002A-treated participants who developed TEAEs compared to placebo
Time Frame: 28 Days
Population: All participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Groups:
- LAM-002A: 71 participants received LAM-002A (Apilimod Dimesylate) 125 mg in five 25-mg capsules BID for 10 days.
- Placebo: 70 participants received Placebo (microcrystalline cellulose) in 5 capsules BID for 10 days.
Arm/Group | LAM-002A | Placebo
Number analyzed (Participants) | 71 | 70
Participants | 26 | 14

3. Secondary Outcome: Clinical Efficacy
Description: Number of Participants with Hospitalization or Death within 28 days
Time Frame: 28 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: 71participants were allocated to receive Placebo (microcrystalline cellulose) in 5 capsules BID for 10 days.
Arm/Group | LAM-002A | Placebo
Number analyzed (Participants) | 71 | 71
Participants
  Yes | 2 | 1
  No | 69 | 70
Statistical Analysis 1: Comparison: LAM-002A vs Placebo; Test type: Superiority — The alternative hypothesis for the statistical testing was that LAM-002A would reduce the cumulative rate of hospitalization or death during the 28-day period comprising 10 days of study drug administration and a further 18 days of observation; p = 0.55, Log Rank; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.18 to 22.89]

4. Secondary Outcome: Change in COVID-19 Clinical Status
Description: To evaluate change in COVID-19 clinical status, as defined by the ordinal scale, of participants treated with LAM-002A compared to placebo at Day 28, in participants who became hospitalized and continued LAM-002A/placebo treatment, based on the following scores:
  1. Not in the hospital
  2. Hospitalized, requiring low flow supplemental oxygen (such as nasal cannula)
  3. Hospitalized, not on invasive ventilation (such as 100% non-rebreather, BIPAP), (pre-ICU)
  4. Hospitalized, in the ICU, on invasive ventilation or Extracorporeal membrane oxygenation (ECMO)
  5. Dead
Time Frame: 28 Days
Population: The intention-to-treat (ITT) population included all participants randomized according to their initial randomized assignment regardless of the treatment actually received.
  * Participant 008-109 in the LAM-002A group was in the hospital at Day 28, but her score is missing, this participant died in the hospital on Day 30.
Measure: Count of Participants; unit: Participants
Arm/Group | LAM-002A | Placebo
Number analyzed (Participants) | 71 | 71
Participants
  1: Not in the hospital | 64 | 66
  2: Hospitalized, requiring low flow supplemental oxygen (such as nasal cannula) | 0 | 0
  3: Hospitalized, not on invasive ventilation (such as 100% non-rebreather, BIPAP), (pre-ICU) | 0 | 0
  4: Hospitalized, in the ICU, on invasive ventilation or ECMO | 0 | 0
  5: Dead | 0 | 0
  Status Unknown* | 7 | 5

5. Secondary Outcome: Oxygen Saturation
Description: Comparison of the number and percentage of participants with an oxygen saturation (O2 sat) ≥95% between LAM-002A versus placebo treatment groups.
Time Frame: Baseline, Day 1, Day 4, Day 11, Day28
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- LAM-002A: 71 participants were allocated to receive LAM-002A (Apilimod Dimesylate) 125 mg in five 25-mg capsules BID for 10 days.nge, Size 0.
Arm/Group | LAM-002A | Placebo
Number analyzed (Participants) | 71 | 71
Participants
  Baseline, oxygen saturation ≥95%: Yes | 67 | 68
  Baseline, oxygen saturation ≥95%: No | 4 | 3
  Day 1, oxygen saturation ≥95%: number analyzed (Participants) | 62 | 61
  Day 1, oxygen saturation ≥95%: Yes | 60 | 59
  Day 1, oxygen saturation ≥95%: No | 2 | 2
  Day 4, oxygen saturation ≥95%: number analyzed (Participants) | 68 | 68
  Day 4, oxygen saturation ≥95%: Yes | 59 | 65
  Day 4, oxygen saturation ≥95%: No | 9 | 3
  Day 11, oxygen saturation ≥95%: number analyzed (Participants) | 64 | 67
  Day 11, oxygen saturation ≥95%: Yes | 60 | 65
  Day 11, oxygen saturation ≥95%: No | 4 | 2
  Day 28, oxygen saturation ≥95%: number analyzed (Participants) | 65 | 66
  Day 28, oxygen saturation ≥95%: Yes | 65 | 66
  Day 28, oxygen saturation ≥95%: No | 0 | 0
Statistical Analysis 1: Comparison: LAM-002A vs Placebo; Risk Difference from generalized estimating equations (GEE) logistic regression at Baseline; Test type: Superiority — The alternative hypothesis for the statistical testing was that a higher proportion of participants would have ≥95% oxygen saturation during LAM-002A administration than during Placebo administration as assessed across Days 1, 4, and 11 of the study drug course; Risk Difference (RD) = -1.4
Statistical Analysis 2: Comparison: LAM-002A vs Placebo; Risk Difference from GEE Logistic Regression at Day 1; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = -1.0
Statistical Analysis 3: Comparison: LAM-002A vs Placebo; Risk Difference from GEE logistic regression at Day 4; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = -8.8
Statistical Analysis 4: Comparison: LAM-002A vs Placebo; Risk Difference from GEE logistic regression at Day 11; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = -3.7

6. Other Pre Specified Outcome: Number and Percentage of Participants With Viral Load < Lower Limit of Quantification (LLOQ)
Description: Evaluated the difference in the number and percentage of participants with a SARS-CoV-2 viral load <LLOQ between the LAM-002A and the placebo arm as measured by a qRT-PCR test from nasopharyngeal samples at Day 4.
Time Frame: 4 Days
Population: Antiviral efficacy population comprising participants with baseline viral load >100,000 copies/ml = log10 viral load >5)
Measure: Count of Participants; unit: Participants
Arm/Group | LAM-002A | Placebo
Number analyzed (Participants) | 37 | 31
Participants | 9 | 3
Statistical Analysis 1: Comparison: LAM-002A vs Placebo; Test type: Superiority — The alternative hypothesis for the statistical testing was that, relative to Placebo, LAM-002A would result in a greater proportion of participants with a SARS-CoV-2 viral load <LLOQ on Day 4; p = 0.20, Fisher Exact — Prespecified significance level of 0.20; Relative Risk = 2.51, 95% CI 2-sided [0.74 to 8.48]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first administration of study drug through Day 28 or when any ongoing drug-related adverse events (AEs) and/or serious adverse events (SAEs) resolved or became stable, up to 30 days.
Description: Adverse Events were analyzed for all participants who received at least 1 dose of study treatment. In the Placebo group, 1 subject did not initiate treatment.
Arm/Group | LAM-002A | Placebo
All-Cause Mortality (participants affected / at risk) | 1/71 | 0/70
Serious Adverse Events (participants affected / at risk) | 2/71 | 1/70
Other Adverse Events (participants affected / at risk) | 26/71 | 15/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAM-002A (N=71) | Placebo (N=70)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAM-002A (N=71) | Placebo (N=70)
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Nausea (Gastrointestinal disorders) | 7 | 3
Vomiting (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Feeling abnormal (General disorders) | 2 | 1
Asthenia (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Chest discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Thirst (General disorders) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 2 | 0
Dizziness postural (Nervous system disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
Respiratory rate increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was potentially limited in its ability to discern a benefit of LAM-002A on viral and clinical endpoints due to the number of participants enrolled, the low baseline viral loads, and the short (4-day) duration of viral load evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agreed that the primary publication, will be coordinated by the sponsor, will be the first publication to present the pooled study results. After the primary publication, or if the primary publication is not published within 2 years of termination of the study, the investigator may freely publish or present the results of his or her work conducted under the clinical trial agreement, subject to providing the sponsor with the opportunity to review the contents.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT04446377/Prot_SAP_000.pdf